CLINICAL TRIAL: NCT02053506
Title: Nutrition Support for Immune Recovery
Brief Title: Nutrition Interventions to Support the Immune System in Response to Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Principal Investigator, Tracey Smith, Research Dietitian, United States Army Research Institute of Environmental Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 13-10-H
Record Dates: First submitted 2014-01-28; First posted 2014-02-03 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Mitigation of Immune Function Decrements in Response to Stress
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immune-enhancing nutritional beverage (Experimental): This group will consume an immune-enhancing beverage and additional protein (1.2-1.5 grams•kg-1 body weight•day-1 versus the RDA of 0.8 grams•kg-1 body weight•day-1) during and after the period of sleep restriction to determine if this nutritional approach attenuate the loss of immune responsiveness.
  Interventions: Dietary Supplement: Immune-enhancing nutritional beverage; Dietary Supplement: Placebo (for nutritional beverage and probiotic)
- Probiotics (BB-12) (Experimental): This group will consume probiotics (BBB12) during and after the period of sleep restriction to determine if nutritional approaches attenuate the loss of immune responsiveness. Consistent with the control group, this group will consume the RDA for protein (0.8 grams•kg-1 body weight•day-1) and placebo beverage (no immune-enhancing vitamins/minerals).
  Interventions: Dietary Supplement: Probiotics (BB-12); Dietary Supplement: Placebo (for nutritional beverage and probiotic)

INTERVENTIONS:
Dietary Supplement: Immune-enhancing nutritional beverage — Combination of arginine, glutamine, omega-3 fatty acids, vitamin C and zinc.
  Arms: Immune-enhancing nutritional beverage
Dietary Supplement: Probiotics (BB-12) — Probiotics (Bifidobacterium Animalis Lactis, BB-12®, Chr Hansen A/S, Hoersholm, Denmark) will be administered as a strawberry-flavored, powdered candy (1 g). The candy will be packaged in a small foil pouch, and each pouch will contain approximately 1 billion colony forming units (CFU) of BB-12® in powder form.
  Other Names: Bifidobacterium Animalis Lactis, BB-12®
  Arms: Probiotics (BB-12)
Dietary Supplement: Placebo (for nutritional beverage and probiotic) — Dietary protein at RDA of 0.8 grams•kg-1 body weight•day-1 and a placebo beverage during and after the period of sleep restriction.

SUMMARY:
Physical and psychological stress on military personnel during training and operational missions can suppress immune function. Creating superficial skin wounds via suction blisters can be used to detect changes in immune function. The goals of this research are to: 1) identify changes in immune function (blood measures and healing time of skin wounds) in response to sleep restriction; and, 2) test the influence of a multi-nutrient beverage and healthy bacteria (i.e., probiotics) on immune function (blood measures and healing time of skin wounds) in response to sleep restriction.

DETAILED DESCRIPTION:
Physical and psychological stress on Warfighters during training and operational missions can suppress immune responsiveness. Skin wound healing models can be used to detect changes in immune function. The goals of this research are to: 1) quantify the impact of an operational stressor (i.e., sleep restriction) on suction blister immune response and skin barrier restoration; and, 2) test the influence of nutrition intervention(s) on immune response and skin barrier restoration consequent to an operational stressor. Research will be conducted in a laboratory environment using male and female Soldiers from the human research participant detachment (NSRDEC), NSRDEC and/or USARIEM. Recently, the investigators lab assessed the test-retest reliability of a suction blister model by creating eight suction blisters on participants' left and right forearms, and sampling blister fluid and skin barrier restoration (12-06H), which will serve as one of the control groups (Group 1, N = 15) for the study described herein. Participants in the study described herein (Groups 2-4, n = ~60) will be exposed to ~50 hours of sleep restriction , after which time eight suction blisters will be induced on one forearm and immune responsiveness and skin barrier restoration time recorded. Participants will receive no nutrition intervention (Group 2), an immune-enhancing beverage and additional protein (1.2 g protein per kg body weight versus 0.8 g protein per kg body weight) (Group 3) or probiotics (Group 4), during and after sleep restriction to determine if nutritional approaches attenuate the loss of immune responsiveness. The results of this study will provide insight into whether nutritional supplementation approaches confer immune recovery. The investigators hypothesize that the suction blister immune response (during the 24 hours following blister induction) and time to skin barrier restoration will degrade after an imposed stress which includes~50 hours of wakefulness and constrained living; and, a diet supplemented with either protein and a multi-nutrient nutritional supplement OR probiotics will attenuate the decrements in suction blister immune responsiveness (during the 24 hours following blister induction) and time to skin barrier restoration in response to ~50 hours of sustained wakefulness and constrained living.

ELIGIBILITY:
Inclusion Criteria:

• Members of the Reserves, National Guard or active duty military personnel

Exclusion Criteria:

* Under the age of 18 or over the age of 45
* Have a tattoo on both forearms
* Are taking nonsteroidal anti-inflammatory drugs (e.g., Advil), aspirin, lipid-lowering drugs or corticosteroids
* Pegnant or lactating
* Imune-compromised (e.g., chemotherapy or radiation treatment)
* Sffering from an autoimmune disease (e.g., lupus)
* Rcovering from a surgery within the past 6 months
* Have an injury that will prevent physical activity
* Have a history of cardiovascular disease
* Are suffering from sleep apnea
* Have a history of psychiatric disorder requiring hospitalization or have taken psychiatric medication (e.g., anti-depressants or anti-anxiety medication) within the past three years for any length of time
* Are suffering from any neurological disorder (e.g., epilepsy or other seizure disorder, narcolepsy or other sleep disorders, or multiple sclerosis)
* Have a BMI ≥ 30.
* Feel uncomfortable handling a weapon, shooting at silhouette targets, ave an injury that will impair firing a rifle
* Have ever been diagnosed with post-traumatic stress disorder
* Are unable to distinguish the color "red" from the color "black".

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2014-01; Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Skin barrier restoration | daily until skin barrier restored (~5-10 days)
  Skin barrier restoration is assessed via transepidermal water loss (TEWL). Skin barrier is considered "restored" when TEWL returns to within 90% of baseline levels.

SECONDARY OUTCOMES:
Suction blister cytokine response | 4, 7 and 24 hours
  Fluid is sampled from blister wound area at various time-points and analyzed for concentration of pro-inflammatory cytokines.

OTHER OUTCOMES:
Leukocyte migration | When blisters are formed (~90 minutes after suction application)
  Leukocyte migration is measured from the blisters after formation and before the top layer of the blister is removed.

CONTACTS AND LOCATIONS:
Overall Officials: Tracey J Smith, PhD, Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- U.S. Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided